CLINICAL TRIAL: NCT02338934
Title: An Open-label Study of Combination of Cinacalcet and Active Vitamin D Analogue in the Management of Severe Secondary Hyperparathyroidism in Haemodialysis Patients
Brief Title: Cinacalcet in Management of Secondary Hyperparathyroidism in Haemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Penang Hospital, Malaysia (Other Government)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr.Ong Loke Meng, Doctor, Penang Hospital, Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT14-HPP-004
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cinacalcet with Vitamin D arm (Experimental): Depending on the iPTH level and the serum calcium level they will be started on Cinacalcet 25mg OD and active Vitamin D will be adjusted. If Serum Cal <2.4 mmol/L - Start Cinacalcet 25mg OD & Increase active Vit D by 1 mcg/dose 3x/week Increase active Vit D by 1 mcg/dose 3x/week or Serum Ca 2.4-2.54 mmol/L- Start Cinacalcet 25mg OD and Maintain active Vit D dose OR if >2.54 mmol/L - Start Cinacalcet 25mg OD & Maintain active Vit D dose. Then they will go to maintenance phase.
  Interventions: Drug: Combination Cinacalcet with Vitamin D analogue

INTERVENTIONS:
Drug: Combination Cinacalcet with Vitamin D analogue — Depending on the iPTH level and the serum calcium level they will be started on Cinacalcet 25mg OD and active Vitamin D will be adjusted. If Serum Cal <2.4 mmol/L - Start Cinacalcet 25mg OD & Increase active Vit D by 1 mcg/dose 3x/week Increase active Vit D by 1 mcg/dose 3x/week or Serum Ca 2.4-2.54 mmol/L- Start Cinacalcet 25mg OD and Maintain active Vit D dose OR if >2.54 mmol/L - Start Cinacalcet 25mg OD & Maintain active Vit D dose. Then they will go to maintenance phase.

SUMMARY:
This is a single arm, open-labelled study to determine the effectiveness of combination Cinacalcet with Vitamin D analogue in the treatment of severe hyperparathyroidism in patients with ESRF on haemodialysis. Patients will be started on PO Cinacalcet 25mg OD + PO/IV active Vitamin D analogues adjusted by increments/decrements in steps of 1 mcg 3x per week every 1-4 weeks until the corrected calcium level is within 2.4-2.54 mmol/L. After iPTH has reached 2-9x ULN, patient enters maintenance phase. If serum calcium falls below 2.1mmol/L, active Vit D dose will be increased and if it is above 2.54 mmol/L, the dose will be decreased.

Percentage reduction of iPTH levels from baseline at 6,12 and 24 months treatment and Percentage of patients achieving iPTH levels within the target range of 2-9x upper limit normal at 6, 12 and 24 months will be determined

DETAILED DESCRIPTION:
Many patients on haemodialysis will develop secondary hyperparathyroidism. Vitamin D analogues such as alphacalcidol are needed to bring their iPTH levels down to normal. However, these analogues can cause hypercalcaemia, thus its doses are limited by this effect. Cinacalcet, which is currently not widely available to patients in hospitals, is a calcimimetic that can reduce both iPTH and serum calcium levels. No studies have yet to be carried out investigating the outcome of using low doses of Cinacalcet as a means of optimizing doses of vitamin D analogues by keeping calcium levels from going over the upper limit. So a single arm, open-labelled study has been designed to determine the effectiveness of combination Cinacalcet with Vitamin D analogue in the treatment of severe hyperparathyroidism in patients with ESRF on haemodialysis. No formal sample size calculation was done as this is a proof of concept study. Power calculation will be done at the end based on the primary outcome of the study.

Methodology: Patients will be started on PO Cinacalcet 25mg OD + PO/IV active Vitamin D analogues adjusted by increments/decrements in steps of 1 mcg 3x per week every 1-4 weeks until the corrected calcium level is within 2.4-2.54 mmol/L. After iPTH has reached 2-9x ULN, patient enters maintenance phase. If serum calcium falls below 2.1mmol/L, active Vit D dose will be increased and if it is above 2.54 mmol/L, the dose will be decreased.

Percentage reduction of iPTH levels from baseline at 6,12 and 24 months treatment and Percentage of patients achieving iPTH levels within the target range of 2-9x upper limit normal at 6, 12 and 24 months will be determined.

ELIGIBILITY:
Inclusion Criteria:1. End Stage Renal Failure (ESRF) patients on haemodialysis with iPTH levels more than 9x upper limit normal 2. Patients who has history of active Vitamin D analogue doses limited by hypercalcaemia (>2.54 mmol/L)

Exclusion Criteria:

1. Pregnant or breastfeeding or planning to become pregnant
2. Life expectancy of 6 months or less
3. History of decompensated liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction of iPTH levels from baseline at 6 months treatment | 6 months

SECONDARY OUTCOMES:
Percentage of patients achieving iPTH levels within the target range of 2-9x upper limit normal at 6, 12 and 24 months | 24 months
The maximum iPTH reduction from baseline | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ong Loke Meng, FRCS, Principal Investigator — Clinical Research Centre, Penang Hospital, Malaysia
Locations (2):
- Malaysia (2):
  - Clinical Research Centre, Penang Hospital, George Town, Pulau Pinang
  - Penang Hospital, George Town, Pulau Pinang